CLINICAL TRIAL: NCT02764671
Title: The Safety and Immunogenicity of 10μg/0.5ml Recombinant Hepatitis B Vaccines(Saccharomyces Cerevisiae) in the Healthy Neonates
Brief Title: Safety and Immunogenicity of Recombinant Hepatitis B Vaccines in the Neonates
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Kangtai Biological Products Co., LTD (Industry)
Collaborators: Guangdong Provincial Institute of Biological Products And Materia Medica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KT0012
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis; Hepatitis B; Liver Diseases; Digestive System Diseases
Keywords: recombinant hepatitis B vaccine; safety; immunogenicity
MeSH Terms: conditions — Hepatitis; Hepatitis B; Liver Diseases; Digestive System Diseases | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 10μg/0.5ml recombinant HBV vaccine (Experimental): 5000 participants who are healthy neonates receive 10μg/0.5ml recombinant hepatitis B vaccine on day 0, 30 and 60.
  Interventions: Biological: 10μg/0.5ml recombinant hepatitis B vaccine

INTERVENTIONS:
Biological: 10μg/0.5ml recombinant hepatitis B vaccine — 5000 participants who are healthy neonates receive 10μg/0.5ml recombinant hepatitis B vaccine on day 0, 30 and 60.

SUMMARY:
The purpose of this study is to further evaluate the immunogenicity and safety of 10μg/0.5ml Recombinant Hepatitis B Vaccines(Saccharomyces Cerevisiae) in the Healthy Neonates.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are healthy full-term infants after birth, Apgar score ≥8;
* Subjects with a birth weight ≥ 2500g;
* Subjects' guardians are able to understand and sign informed consent;
* Subjects who can and will comply with the requirements of the protocol.

Exclusion Criteria:

* Family history of eclampsia, epilepsy and encephalopathy;
* Subjects' birth mother had immune system dysfunction, or history of organ transplantation or blood dialysis;
* Subjects' parents had a medical history of allergic to any ingredient of the vaccine, including supplementary material and formaldehyde;
* Subjects' parents had a medical history of allergic to combined hepatitis A and B vaccine(HAB) or hepatitis B vaccine;
* Subjects had serious acute and chronic diseases;
* with temperature ≧37.1℃;
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives.

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5000 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Within 30 days after hepatitis B vaccination

SECONDARY OUTCOMES:
Geometric mean titer of anti-hepatitis B virus surface antigen antibody | The 30th day after whole course of hepatitis B vaccination
  Geometric mean titer of anti-hepatitis B virus surface antigen antibody was measured by chemiluminescence assay and expressed with mIU/mL.
Geometric mean titer of anti-hepatitis B virus surface antigen antibody | The 1th year after whole course of hepatitis B vaccination
  Geometric mean titer of anti-hepatitis B virus surface antigen antibody was measured by chemiluminescence assay and expressed with mIU/mL.
Geometric mean titer of anti-hepatitis B virus surface antigen antibody | The 2th year after whole course of hepatitis B vaccination
  Geometric mean titer of anti-hepatitis B virus surface antigen antibody was measured by chemiluminescence assay and expressed with mIU/mL.
Geometric mean titer of anti-hepatitis B virus surface antigen antibody | The 3th year after whole course of hepatitis B vaccination
  Geometric mean titer of anti-hepatitis B virus surface antigen antibody was measured by chemiluminescence assay and expressed with mIU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Huizhen, master, Principal Investigator — Guangdong Center for Disease Prevention and Control
Locations (2):
- China (2):
  - Gaozhou District Center for Disease Control and Prevention, Maoming, Guangdong
  - Xinxing District Center for Disease Control and Prevention, Yunfu, Guangdong